CLINICAL TRIAL: NCT01408602
Title: A 24-week, Phase 2, Double-blind, Placebo-controlled, Randomized Study to Assess the Safety and Efficacy of 2 Doses of MRC375 in Patients With Moderate to Severe Rheumatoid Arthritis
Brief Title: A Study of Two Doses of MRC375 in Moderate to Severe Rheumatoid Arthritis Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Molecular Research Center, Inc. (Industry)
Collaborators: Camargo Pharmaceutical Services (Industry); Clin Data Services (Unknown); Harrison Clinical Research (Industry); BARC Global Central Laboratory (Unknown); Bilcare Global Clinical Supplies (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MRC2011-001
Record Dates: First submitted 2011-08-02; First posted 2011-08-03 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- MRC375 75 mg (Experimental): MRC375 (enteric coated Tetracycline) 75 mg 3 times a day
  Interventions: Drug: MRC375
- MRC375 150mg (Experimental): MRC375 (enteric coated Tetracycline) 150mg 3 times a day for 24 weeks.
  Interventions: Drug: MRC375 150mg
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: MRC375 — MRC 375 (enteric coated Tetracycline) 75mg 3 times a day for 24 weeks.
  Arms: MRC375 75 mg
Drug: Matching Placebo — Matching Placebo 3 times a day for 24 weeks. Early escape at week 16,20.
  Arms: Placebo
Drug: MRC375 150mg — MRC375 (enteric coated Tetracycline) 150mg 3 times a day for 24 weeks
  Arms: MRC375 150mg

SUMMARY:
This study will treat moderate to severe rheumatoid arthritis with MRC375 (either 75 mg 3 times a day, 150 mg 3 times a day or placebo 3 times a day)in patients 18 years of age or older that can be currently on low doses of methotrexate or can stop treatment of current RA medications to enter the study. Safety of MRC375 will also be evaluated. There are up to 8 clinic visits over 24 weeks.

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled study to assess the safety and efficacy of MRC375 at 75 mg or 150 mg with matching placebo (taken tid with meal or light snack) in patients with moderate to severe RA. Patients will be randomized to one of the following study arms for 24 weeks:

* Treatment 1, Placebo: 2 tablets taken tid
* Treatment 2, MRC375: 1 tablet of 75 mg tetracycline HCL plus 1 matching placebo tablet taken tid. Total daily dose = 225 mg.
* Treatment 3, MRC375: 2 tablets of 75 mg tetracycline HCL taken tid. Total daily dose = 450 mg.

Study medication should be taken within 30 minutes of a meal or light snack (either before or after).

ELIGIBILITY:
Inclusion Criteria:

1. Is 18 years of age
2. Is diagnosed with moderate to severe adult onset RA > = 6 months duration, as defined by the 1987 ACR classification criteria
3. Has moderate to severe RA as defined by:

   * ≥4 tender joints/painful (28 joint count) at screening
   * ≥4 swollen joints (28 joint count) at screening
4. Has a Health Assessment Questionnaire (HAQ) of >0
5. Has a physician global assessment (Likert scale) of >0
6. Has a patient global assessment of pain (Likert scale) of >0
7. Has a patient assessment of pain (Likert scale) of >0
8. Has stable doses of the following allowable medications during the study, if applicable:

   * Stable dose of NSAIDs or other analgesics for at least 2 weeks prior to administration of study drug at regulatory approved doses
   * Stable dose of methotrexate 7.5 mg to 25 mg/day once weekly for at least 6 weeks prior to administration of study drug (no changes in dosing regimen for 4 weeks prior to screening)
   * Stable dose of hydroxychloroquine either monotherapy or in combination with methotrexate 8 weeks prior to administration of study drug
9. Is a non-pregnant, non-lactating female who is postmenopausal, naturally or surgically sterile, or who agree to use effective contraceptive methods throughout the course of the study. Postmenopausal is defined as at least 12 months natural spontaneous amenorrhea
10. If female of childbearing potential, must agree to use one of the following acceptable birth control methods:

    * Surgically sterile (bilateral tubal ligation with surgery at least 6 weeks prior to screening, hysterectomy, or bilateral oophorectomy);
    * Intrauterine device (IUD) in place for at least 3 months prior to first dose of study drug;
    * Abstinence (not having sexual intercourse);
    * Barrier method (condom or diaphragm) with spermicide for at least 14 days prior to screening and through study completion;
    * Stable hormonal contraceptive for at least 3 months prior to study and through study completion
11. If female of childbearing potential, has a negative serum hCG pregnancy test at screening
12. Is able to swallow whole tablets of orally administered medication
13. Is able to understand and provide signed informed consent.

Exclusion Criteria:

1. Has been diagnosed with any other inflammatory arthritis (eg, psoriatic arthritis)
2. Has a secondary type of arthritis (eg, osteoarthritis) that would interfere with study evaluations
3. Has taken the following drugs within the timeframe specified below:

   * Infliximab, etanercept, adalimumab, abatacept, or other biological therapies (except rituximab) - Within 12 weeks prior to the administration of study drug;
   * Rituximab - Within 12 months prior to the administration of study drug;
   * Disease-modifying antirheumatic drugs (DMARDs) or other anti-rheumatic therapies not specified above including but not limited to: sulfasalazine, gold, leflunomide, penicillamine, dapsone, azathioprine, 6-mercaptopurine, chlorambucil, cyclophosphamide, cyclosporin, mycophenolate mofetil - Within 12 weeks prior to the administration of study drug;
   * Any steroids (glucocorticoids); glucocorticoids must be discontinued for at least 4 weeks prior to administration of study drug. Intraarticular, intramuscular, or intravenous glucocorticoids must not have been given at least 6 weeks prior to administration of study drug.
   * Note: Use of probiotics is allowed and is NOT an exclusion criterion.
4. Has a uncontrolled symptoms of fibromyalgia with sufficient symptoms requiring treatment (NOTE: patients on a stable dose of treatment for symptoms of fibromyalgia ≥ 4 weeks will be allowed in the study.)
5. Has a history of allergic reaction to tetracycline or other related drugs
6. Had major surgery or trauma within 28 days prior to screening
7. Is concurrently using minocycline or doxycycline (washout of 4 weeks required before the administration of study drug)
8. Patients who are on chronic antibiotics or who are on antibiotics for GI infections (such as Clostridium difficile)
9. Has clinically significant ECG abnormalities
10. Has any clinically significant abnormal laboratory test results found during medical screening including: AST or ALT > 2 x upper limit of normal or serum creatinine > 2.0 mg/dL
11. Has clinically significant history or presence of any gastrointestinal pathology (eg, chronic diarrhea, inflammatory bowel disease, acute diverticulitis), irritable bowel syndrome, unresolved gastrointestinal symptoms (eg. diarrhea, vomiting, symptoms of acute diverticulitis), liver or kidney disease, gastric bypass, gastric stapling, use of Lap-Band®, or other conditions known to or which might interfere with the absorption, distribution, metabolism, or excretion of the drug
12. Has any historical or active neurological, endocrine, cardiovascular, pulmonary, hematological, psychiatric, or metabolic disease that is considered clinically significant by the Investigator
13. Has known history of HIV, hepatitis B or C (patients that have positive hepatitis B serology due to prior vaccination will be allowed in the study)
14. Has an active malignancy of any type or history of malignancy. Patients who have a history of a successfully treated non-metastatic cutaneous squamous cell or basal cell carcinoma (ie. non melanoma skin cancer)and/or localized carcinoma in situ of the cervix are eligible. Patients with a history of other malignancies that have been treated and who have no evidence of recurrence for at least 5 years before study enrollment are also eligible.
15. Has difficulty swallowing tablets
16. Is ACR Functional Class IV (limited ability to perform usual self-care, vocational, and avocational activities)
17. Has known or suspected pregnancy, planned pregnancy, or lactation (for female patients)
18. Has clinically significant mental illness (to be determined by the Investigator)
19. Has a history in the last 2 years or current evidence of abuse of illicit drugs, prescription medications, or alcohol that, in the opinion of the Investigator, would interfere with adherence to study requirements. Has exposure to any investigational agent within 30 days prior to study entry.
20. Was previously enrolled in this study
21. Has recent history of bacterial intestinal tract infection (gastroenteritis, colitis, diverticulitis, appendicitis)
22. Has a condition the Investigator believes would interfere with the ability to provide informed consent or comply with study instructions, or that might confound the interpretation of the study results or put the patient at undue risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2011-11; Primary Completion 2014-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Efficacy evaluated of both doses of MRC375 compared to placebo after 24 weeks of treatment as measured by the rate of achievement of 20% improvement in ACR criteria | 24 weeks
  evaluate efficacy of both doses of MRC375 compared to placebo after 24 weeks of treatment, as measured by a rate of achievement of 20% improvement in American College of Rheumatology (ACR) criteria (ACR20) at Week 24

SECONDARY OUTCOMES:
Safety and tolerability of both doses of MRC375 | 24 weeks
  evaluate the safety and tolerability of both doses of MRC375 tablets
Compare the Efficacy of two doses of MRC375 when compared to a placebo for the change from baseline screening in each of the individual ACR components measuring RA after 24 weeks of treatment | 24 weeks
  compare the efficacy of 2 doses of MRC375 tablets (75 mg tid and 150 mg tid) when compared to placebo for the change from baseline screening in each of the individual ACR components measuring rheumatoid arthritis (RA) after 24 weeks of treatment.

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Mobile Diagnostic Center Rheumatology, Mobile, Alabama
  - Valerius Medical Group, Long Beach, California
  - Trial Concierge/Pacific Clinical Studies, Los Alamitos, California
  - Axis Clinical Trials, Los Angeles, California
  - Riverside Clinical Research, Edgewater, Florida
  - Global Clinical Professionals, Miami, Florida
  - The Arthritis Center, Palm Harbor, Florida
  - Lakeview Medical Research, Summerfield, Florida
  - Analan Clinical Research, Lenexa, Kansas
  - Trial Concierge, Owensboro, Kentucky
  - Quality Clinical Research, Inc., Omaha, Nebraska
  - Advanced BioMedical Research of America, Las Vegas, Nevada
  - Arthritis Center of Reno, Reno, Nevada
  - PMG Research of Salisbury, Salisbury, North Carolina
  - Providence Health Partners, Dayton, Ohio
  - Paramount Medical Research & Consulting, LLC, Middleburg Heights, Ohio
  - The Center for Excellence in Aging and Geriatric Health, Williamsburg, Virginia
  - Apex Clinical Research, Kennewick, Washington
  - South Puget Sound Clinical Research Center, Olympia, Washington